CLINICAL TRIAL: NCT03953781
Title: Effect of Valproate Versus Levetiracetam Monotherapy on Reproductive Functions in Newly Diagnosed Epileptic Males
Brief Title: Effect of Valproate Versus Levetiracetam Monotherapy on Reproductive Functions in Epileptic Males
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, rania sanad, Principal Investigator, Zagazig University
Other Study IDs: ZU-IRB#4731\ 24-1-2018
Record Dates: First submitted 2019-04-17; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; antiepileptic drugs; males; reproduction
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: 25 participants, were treated by valproate (VPA) as a monotherapy till became seizure free at the last 8-weeks before post treatment check-point, with ages ranged from 18-43 years
  Interventions: Drug: Effect of valporate on Reproductive Functions in Newly Diagnosed Epileptic Males
- group 2: 25 participants were treated by levetiracetam (LEV) with the same regimens of valproate as a monotherapy, with ages ranged from 20-45 years.
  Interventions: Drug: Effect of levetiracetam on epileptic males reproductive function

INTERVENTIONS:
Drug: Effect of valporate on Reproductive Functions in Newly Diagnosed Epileptic Males
  Other Names: Effect of depakin monotherapy on epileptic males reproductive function
  Groups: group 1
Drug: Effect of levetiracetam on epileptic males reproductive function
  Other Names: Effect of levepex on epileptic males reproductive function
  Groups: group 2

SUMMARY:
Background: Different antiepileptic drugs are responsible for reproductive dysfunction in male epileptic patients. The aim of this study is to evaluate the effect of valproate versus levetiracetam as a monotherapy on males' sex hormones and sperm parameters in newly diagnosed epilepsy. Methods: This comparative study included 50 newly diagnosed epileptic male participants from outpatient clinic of Neurology department of Zagazig University Hospitals. All participants were subjected to complete general and neurological examination, Doppler ultrasonography of the testis, pre and post treatment serum sex hormone assay and semen analysis. Post- treatment re- evaluation check point was determined if eight weeks have passed after the last seizures. This study included two groups, group I: 25 participants, were treated by valproate (VPA) as a monotherapy till became seizure free at the last 8-weeks before post treatment check-point, with ages ranged from 18-43 years. Group II: 25 participants were treated by levetiracetam (LEV) with the same regimens of valproate as a monotherapy, with ages ranged from 20-45 years.

DETAILED DESCRIPTION:
Background: Epilepsy is a chronic neurological disorder characterized by recurrent epileptic attacks and researches have reported that the relation between epilepsy and the reproductive dysfunction is not yet completely understood. Seizures are linked with sexual dysfunction as part of the disease pathophysiology in these patients. Through epileptic discharge, hypothalamus receives signals from hippocampus, amygdala and cerebral cortex. Hypothalamic-pituitary axis signaling changes is leading to sex hormones release including follicle stimulating hormones and luteinizing hormone changes.

However, the available antiepileptic drugs (AED) have not yet been proven to have negative impacts on sexual function. Evaluation of AED induced sexual dysfunction is complicated, less than clear, and is hard to find. Sex hormone levels can be changed due to AEDs which are the cause of sexual dysfunction and reproductive disorders Different antiepileptic drugs are responsible for reproductive dysfunction in male epileptic patients. The aim of this study is to evaluate the effect of valproate versus levetiracetam as a monotherapy on males' sex hormones and sperm parameters in newly diagnosed epilepsy. Methods: This comparative study included 50 newly diagnosed epileptic male participants from outpatient clinic of Neurology department of Zagazig University Hospitals. All participants were subjected to complete general and neurological examination, Doppler ultrasonography of the testis, pre and post treatment serum sex hormone assay and semen analysis. Post- treatment re- evaluation check point was determined if eight weeks have passed after the last seizures. This study included two groups, group I: 25 participants, were treated by valproate (VPA) as a monotherapy till became seizure free at the last 8-weeks before post treatment check-point, with ages ranged from 18-43 years. Group II: 25 participants were treated by levetiracetam (LEV) with the same regimens of valproate as a monotherapy, with ages ranged from 20-45 years.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-45 years.
* All participants had normal brain imaging (Brain CT or MRI).
* All participants had normal thyroid functions and normal sex hormones assay.

Exclusion Criteria:

* participants are currently receiving hormonal replacement therapy, or any drugs that may affect reproductive functions were excluded.
* participants with significant or progressive medical illness.
* participants with testicular atrophy, varicocele or infectious diseases .

Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study included 50 newly diagnosed epileptic males (clinically and electro physiologically ((EEG)) according to the International League against Epilepsy ((ILAE)) classification 2010)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
the effect of valproate on males' sex hormones in newly diagnosed epileptic males. | 8-weeks
  percent of valproate treated patients with change in luteinizing hormone and follicle stimulating hormones and prolactin serum level.
the effect of valproate on sperm parameters in newly diagnosed epileptic males. | 8-weeks
  percent of valproate treated patients with change in semen analysis parameters.
the effect of levetiracetam on males' sex hormones in newly diagnosed epileptic males. | 8-weeks
  percent of levetiracetam treated patients with change in luteinizing hormone and follicle stimulating hormones and prolactin serum level.
the effect of levetiracetam on sperm parameters in newly diagnosed epileptic males. | 8-weeks
  percent of levetiracetam treated patients with change in semen analysis parameters.

IPD SHARING:
Plan to Share IPD: Yes
after publishing the manuscript in the Egyptian journal of neurology, psychiatry and neurosurgery
Supporting Information: Study Protocol, SAP
Time Frame: after publishing the manuscript in the Egyptian journal of neurology, psychiatry and neurosurgery
Access Criteria: after publishing the manuscript in the Egyptian journal of neurology, psychiatry and neurosurgery
URL: http://ejnpn.springeropen.com